CLINICAL TRIAL: NCT06760091
Title: Multicentric Registry Study of Autoimmune Encephalitis
Brief Title: A Multicentric Cohort of Autoimmune Encephalitis
Status: Not yet recruiting | Type: Observational
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Other Study IDs: XMEC-2024-003
Record Dates: First submitted 2024-12-30; First posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-12

CONDITIONS: Autoimmune Encephalitis
MeSH Terms: conditions — Autoimmune Diseases of the Nervous System

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The biological samples of enrolled patients, such as blood, cerebrospinal fluid and teratoma samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- autoimmune encephalitis group
  Interventions: Other: baseline data collection and follow-up

INTERVENTIONS:
Other: baseline data collection and follow-up — At the time of enrollment, baseline characteristics will be collected, and each subject will be followed up for 2 years through face-to-face, telephone, or online visits. During the follow-up period, the clinical prognosis will be recorded.

SUMMARY:
This study aims to establish an autoimmune encephalitis cohort and observe the prognosis of patients with different subtypes and subgroups (e.g. epilepsy subgroup and teratoma subgroup ). Clinical characteristics, biological samples, and imaging data will be collected to discover blood and imaging biomarkers for providing support for the treatment, early warning, and outcome prediction.

ELIGIBILITY:
Inclusion Criteria:

* 1. Gender and age are not limited; 2. Newly diagnosed autoimmune encephalitis according to at least one of the following three criteria:

  1. According to the criteria of Graus et al in 2016, diagnosed as "definite autoimmune limbic encephalitis"
  2. According to the criteria of Graus et al in 2016, diagnosed as "possible autoimmune encephalitis" and typical autoantibodies are detected in serum or cerebrospinal fluid
  3. According to the criteria of Graus et al in 2021, diagnosed as "possible or definite paraneoplastic neurological syndrome" (excluding peripheral nervous system syndrome) 3. The patient or legal representative voluntarily signed the paper informed consent form.

Additional inclusion criteria for patients in the epilepsy subgroup: patients diagnosed with epilepsy secondary to autoimmune encephalitis.

Exclusion Criteria:

* No additional exclusion criteria

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with autoimmune encephalitis or paraneoplastic neurological syndrome will be enrolled and no additional exclusion criteria are set.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-02-01 (Estimated); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in modified Rankin score (mRS) from baseline | 3months, 6 months, 12months, 24months
  Change in modified Rankin score (mRS) from baseline at month 1, month 3, month 6(mRS : Minimum Score 0, Maximum score 6, higher scores mean a worse outcome).

SECONDARY OUTCOMES:
Proportion of Subjects With Occurrence | 12 months, 24 months
Change of Clinical Assessment Scale in Autoimmune Encephalitis (CASE) Score from Baseline | 3months, 6 months, 12months, 24months
  The Clinical Assessment Scale in Autoimmune Encephalitis (CASE) score is designed specifically to assess the severity of autoimmune disease. It is a general scoring system ranging from 0 to 27 and can be used as an alternative tool to assess the severity of patients with AE more accurately. Higher scores mean a worse clinical status.
Changes of pathogenic antibody titers from baseline | 3months, 6 months, 12months, 24months

CONTACTS AND LOCATIONS:
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, China

IPD SHARING:
Plan to Share IPD: No